CLINICAL TRIAL: NCT02053597
Title: A Phase II TRIal evalUating the Menstrual and Ovarian Function of Young Breast Cancer Patients Treated With a cycloPHosphamide-free Regimen Composed of Doxorubicin and Paclitaxel
Brief Title: TRIal evalUating the Menstrual and Ovarian Function of Young Breast Cancer Patients Treated With a cycloPHosphamide-free Regimen
Acronym: TRIUMPH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: due to evolving scientific knowledge in the field that would make the questions being addressed in the trial less relevant
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE2142; 2013-000173-77 (EudraCT Number)
Record Dates: First submitted 2014-01-27; First posted 2014-02-03 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Primary breast cancer; Young women; Ovarian function; Sexual function; Eligible for adjuvant or neoadjuvant chemotherapy; Negative hormone-receptor status
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- doxorubicin and paclitaxel (Experimental): All patients will receive four cycles of doxorubicin (A) (50 mg/m2) and paclitaxel (P) (200 mg/m2), given on a three-weekly basis for four cycles, followed by weekly paclitaxel (P) (80 mg/m2) for twelve weeks.
  Interventions: Drug: Doxorubicin; Drug: paclitaxel

INTERVENTIONS:
Drug: Doxorubicin — All patients will receive four cycles of doxorubicin (A) (50 mg/m2)
Drug: paclitaxel — All patients will receive four cycles paclitaxel (P) (200 mg/m2), given on a three-weekly basis for four cycles, followed by weekly paclitaxel (P) (80 mg/m2) for twelve weeks.

SUMMARY:
Recently, there has been a rising trend of delaying childbearing and hence more women are diagnosed with breast cancer before completing their families. Given the continuous decline in recurrences and death secondary to breast cancer and the reassuring data on the safety of pregnancy following breast cancer more women are inquiring into the possibility of preserving fertility following chemotherapy. The challenge remains in using a regimen that is devoid of cyclophosphamide, but is as effective as the standard regimens that incorporate cyclophosphamide. The combination doxorubicin (50 mg/m2) and paclitaxel (200 mg/m2) (AP) followed by 12 weeks of paclitaxel (80 mg/m2) (P) emerges as a treatment option with convincing results regarding its effectiveness in the early setting, and could be potentially associated with less ovarian toxicity being devoid of cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 40 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
3. Non-metastatic primary invasive carcinoma of the breast eligible for adjuvant or neoadjuvant chemotherapy.
4. Negative estrogen (ER) and progesterone receptor (PgR) status.
5. Baseline left ventricular ejection fraction (LVEF) ≥50% measured by an echocardiogram or MUGA.
6. Interested in maintaining menstrual and/or ovarian function following completion of chemotherapy.
7. Known HER2/neu status.
8. Negative pregnancy test within 14 days prior to starting chemotherapy.
9. Adequate hematologic, hepatic and renal function.
10. Signed informed consent.

Exclusion Criteria:

1. History of prior malignant disease (breast or non-breast) or non-malignant condition which was treated with chemotherapy, pelvic irradiation or any therapy that could potentially affect ovarian function.
2. Previous history of amenorrhea > 3 months within the last 2 years (excluding pregnancy).
3. Ovarian insufficiency defined as serum FSH > 20 IU/L at the local laboratory, anytime during the menstrual cycle.
4. Any ovarian pathology or abnormalities at the screening pelvic ultrasound, except for functional follicular cysts.
5. Pregnant or breastfeeding patients.
6. Inability or unwillingness to use effective contraception during and up to 3 months after the last dose of study medication. Effective methods include the following: non-hormonal intrauterine device, barrier method - condoms, diaphragm - also in conjugation with spermicidal jelly, or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed.
7. Concurrent use of any other cytotoxic or hormonal agent, namely GnRH agonists.
8. Prior pre-existing peripheral neuropathy of any cause, including diabetes mellitus, alcohol abuse, HIV infection, autoimmune and hereditary neuropathies, amyloidosis, hypothyroidism, vitamin deficiencies.
9. Serious cardiac illness, uncontrolled hypertension or medical condition that would affect administration of chemotherapy and compliance to study procedures.
10. Known sensitivity to any of the study medications.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ovarian function | At screening, after 4 cycles of chemotherapy, at the end of chemotherapy, at 6, 12, 18 and 24 months following chemotherapy
  Ovarian function will be evaluated using serum FSH, estradiol and AMH. Ovarian failure is defined as serum FSH >40 IU/L. Ovarian insufficiency is defined as serum FSH level from 20 - 40 IU/L. Ovarian reserve will be evaluated by serum AMH. Adequate ovarian reserve is defined as serum AMH >1 ng/ml. Menstrual function will be evaluated by collecting information of the 1st day of last menstrual cycle, and cycle length (days between two menstruating periods).
  Ovarian function will be evaluated using serum FSH, estradiol and AMH. Ovarian failure is defined as serum FSH >40 IU/L. Ovarian insufficiency is defined as serum FSH level from 20 - 40 IU/L. Ovarian reserve will be evaluated by serum AMH. Adequate ovarian reserve is defined as serum AMH >1 ng/ml.
Change from baseline in menstrual function | At screening, after 4 cycles of chemotherapy, at the end of chemotherapy, at 6, 12, 18 and 24 months following chemotherapy
  Menstrual function will be evaluated by collecting information of the 1st day of last menstrual cycle, and cycle length (days between two menstruating periods). In patients menstruating regularly after 12 months of chemotherapy cessation, information on menstrual cycle will be collected at 6-monthly intervals until developing menopause, disease recurrence, becoming pregnant, whichever occurs earlier, for a maximum period of 5 years after end of chemotherapy.

SECONDARY OUTCOMES:
Ovarian reserve | At 12 months following the end of chemotherapy.
  A serum AMH determination will be performed at 12 months after the end of chemotherapy. An adequate ovarian reserve is defined as serum AMH >1 ng/ml at that timepoint.
Occurence of Adverse Events | From the signature of informed consent until until the end of study treatment/treatment discontinuation visit 30 days after the last dose of study medication
  This study will use the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0, for adverse event reporting.
Impact of treatment on the behavior of menstruation after menses resumption | At 18, 24 and 60 months after end of chemotherapy.
  In patients menstruating regularly after 12 months of chemotherapy cessation, information on menstrual cycles will be collected at 18, 24 and up to 60 months after end of chemotherapy, until developing menopause, disease recurrence or becoming pregnant, whichever occurs earlier. This information will include the date of last menstrual period, menstruation duration and if 2 or more consecutive menstrual cycles were missed, allowing to assess irregularity and possible cessation of menses.
Evaluate the impact of a cyclophosphamide-free regimen on sexual function | At baseline, after 4 cycles, end of chemotherapy, 6, 12 and 24 months following the end of chemotherapy.
  Patient will complete two validated health-related quality of life questionnaires, one on menopausal symptoms (FACT-ES version 4) and the other on sexual functioning (FSAQ).
Evaluate the impact of the regimen on peripheral neurotoxicity | At baseline, after 4 cycles, end of chemotherapy, 6, 12 and 24 months following the end of chemotherapy.
  Patient will complete one validated health-related quality of life questionnaire on peripheral neurotoxicity (FACT-Taxane version 4).
Pregnancy rate after cessation of chemotherapy | From end of chemotherapy up until 60 months after.
  Number of pregnancies among participants.
Event-free survival | From the date of registration up until 60 months after the end of chemotherapy.
  Event-free survival will be calculated from the date of registration to the study to developing local, loco-regional or distant metastasis, secondary malignancies or death. All patients will be considered for the primary efficacy analysis (ITT analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Daphné Tkint de Roodenbeke, MD, PhD, Principal Investigator — Jules Bordet Institute; Hatem Azim, MD, PhD, Principal Investigator — Jules Bordet Institute; Isabelle Demeestere, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (4):
- Belgium (4):
  - Jules Bordet Institute, Brussels, Brussels Capital
  - Hôpital Erasme, Brussels, Brussels Capital
  - Clinique et Maternité Sainte Elisabeth, Namur, Namur
  - GZA Ziekenhuisen Campus Sint-Augustinus - Iridium Kankernetwerk, Antwerp, Wilrijk